CLINICAL TRIAL: NCT00959101
Title: A Randomised, Single-Blind, Three-Period Crossover Study Examining the Single Dose Pharmacokinetics of Concomitantly Administered Repaglinide and Metformin Versus Combination Tablet Dosing (NN4440) in Fed Healthy Male Volunteers
Brief Title: Comparison of Repaglinide and Metformin Combination Tablet Versus Repaglinide and Metformin as Separate Tablets in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NN4440-1963
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — repaglinide; Metformin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental)
  Interventions: Drug: repaglinide and metformin combination tablet
- B (Experimental)
  Interventions: Drug: repaglinide and metformin combination tablet
- C (Active Comparator)
  Interventions: Drug: repaglinide; Drug: metformin

INTERVENTIONS:
Drug: repaglinide and metformin combination tablet — Combination tablet of repaglinide (1.0 mg)/metformin (500 mg) given just prior to a standard normal breakfast
  Arms: A
Drug: repaglinide and metformin combination tablet — Combination tablet of repaglinide (2.0 mg)/metformin (500 mg) given just prior to a standard normal breakfast
  Arms: B
Drug: repaglinide — Co-administration of metformin 500 mg tablet and repaglinide 2 mg tablet given just prior to a standard normal breakfast
  Arms: C
Drug: metformin — Concomitant administration: Metformin 500 mg tablet and Repaglinide 2 mg tablet
  Arms: C

SUMMARY:
This trial is conducted in Asia. The aim of this clinical trial is to investigate the bioequivalence of repaglinide and metformin combination tablet versus repaglinide and metformin as coadministered tablets after meal.

The trial is designed as a three-period, six-sequence, single-dose, crossover pharmacokinetic trial where the trial participant is randomised to one of six possible treatment periods (Williams design). The trial participant will receive one single dose of each trial product in varying order.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign informed consent before initiating any trial related procedures
* BMI: 19.0-25.0 kg/m2
* Fasting plasma glucose: 3.9-6.1 mmol/L
* Trial participant is judged to be in good health on the basis of their medical history, physical examination, ECG, and routine laboratory data

Exclusion Criteria:

* Any clinically significant disease history, in the opinion of the Investigator, of systemic or organ disease
* Clinically significant abnormalities on pre-study clinical examination or any laboratory measurements during screening
* Any regular use of prescription or nonprescription drugs, including mega-vitamin or herbal supplement regimens that cannot be stopped at least two weeks prior to start of treatment and for the duration of the trial
* Currently a smoker (more than one cigarette per day or equivalent)
* Use of grapefruit or grapefruit juice within 7 days of trial product dose administration
* Blood donation, surgery or trauma with significant blood loss (400 mL) within the last 2 months prior to trial product dose administration
* Recent history (within the last 2 years) of drug or alcohol abuse
* Known or suspected allergy to trial product or any of the excipients or a history of multiple and/or severe allergies to drugs or foods or of severe anaphylactic reactions
* Subject has taken an investigational drug in another clinical trial within the last 4 weeks.
* Recent history (within the last 3 month) of nausea, diarrhea or gastrointestinal complaints
* History of any illness that, in the opinion of the Investigator, might confound the results of the trial or pose additional risk in administering trial product to the trial participant

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
AUC0-t and Cmax (after repaglinide 2.0 mg and metformin 500 mg as co-administered tablets and combination tablet dosing under fed state) | 24hr profile after single dose of trial drug in each treatment period

SECONDARY OUTCOMES:
Repaglinide AUC(0-24 & 0-∞) and Cmax after combination tablet (repaglinide 1.0 mg/metformin 500 mg) during fed state | 24hr profile after single dose of trial drug in each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Beijing, Beijing Municipality, China

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com